CLINICAL TRIAL: NCT06245629
Title: Bortezomib-bendamustine-melphalan vs High-dose Melphalan in Autologous Hematopoietic Stem Cell Transplantation for Relapsed Multiple Myeloma - a Single Center Retrospective Cohort Study
Brief Title: Bortezomib-bendamustine-melphalan vs Melphalan for Multiple Myeloma
Status: Recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Uppsala County Council, Sweden (Other Government); Dalarna County Council, Sweden (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-04134-01
Record Dates: First submitted 2023-09-26; First posted 2024-02-07 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Myeloma Multiple
Keywords: Autologous hematopoietic stem cell transplantation; Melphalan; Bendamustine; Bortezomib
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Bortezomib-bendamustine-melphalan: Myeloma patients receiving bortezomib-bendamustine-melphalan at autologous hematopoietic stem cell transplantation first relapse.
  Interventions: Drug: Bortezomib-bendamustine-melphalan
- high-dose melphalan: Myeloma patients receiving high-dose melphalan at autologous hematopoietic stem cell transplantation at first relapse.

INTERVENTIONS:
Drug: Bortezomib-bendamustine-melphalan — The aim of this retrospective cohort study is to evaluate the efficacy and safety of the conditioning regimen BBM compared to HDM in the setting of relapsed multiple myeloma.
  Other Names: High-dose melphalan
  Groups: Bortezomib-bendamustine-melphalan

SUMMARY:
This project will evaluate the efficacy and safety of the conditioning regimen bortezomib-bendamustine-melphalan (BBM) in combination with autologous hematopoietic stem cell transplantation (ASCT) in relapsed multiple myeloma given from 2011 to 2018 at Uppsala University Hospital. This approach will be retrospectively compared to high dose melphalan (HDM) in the same setting in the years prior to, and following the BBM-period. Data on efficacy and safety data will be collected through systematic analysis of electronic medical records and from the Swedish Cancer Registry.

DETAILED DESCRIPTION:
Study design This is a retrospective single center cohort study comparing the new conditioning regimen bortezomib-bendamustine-melphalan to standard high-dose melphalan. The data sources will be electronic medical records and prospectively collected data from the Swedish Cancer Registry. The comparison will be analyzed in two parts. First, each patient will be its own control, comparing time to next treatment (TNT) for the first ASCT (always HDM, referred to as ASCT1) and second ASCT (BBM or HDM, referred to as ASCT2), and compare the mean difference between the two cohorts. Secondly, the difference in efficacy and severe adverse events between BBM and HDM at ASCT2 will be compared.

Study population Fifty consecutive patients, who were referred to Uppsala University Hospital (UUH) for a second ASCT after relapse in multiple myeloma following HDM and ASCT between 1 Nov 2011 and 30 Oct 2018 and who received conditioning with bortezomib-bendamustine-melphalan will be included in this study. As a control group, 25 consecutive patients who were treated with HDM prior to 1 Nov 2011 and 25 consecutive patients following 30 Oct 2018. The patients will be identified through the local European Society for Blood and Marrow Transplantation (EBMT) registry at UUH.

UUH is the referral hospital for seven Swedish regions with a total population of 2 151 353 at Dec 31 2022, which constitutes roughly one fifth of the population of Sweden.

Data collection Study data will be collected through systematic analysis of medical records from UUH and all the hospitals referring patients to UUH and from the Swedish Cancer Registry. All severe adverse events (AEs) will be collected until day 100 after ASCT2 according to National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

Primary endpoints

• Mean TNT after ASCT1 and ASCT2 for each individual patient (each patient as its own control), for BBM and HDM-treated patients

Secondary endpoints

* Median time to next treatment (TNT) after ASCT2
* Median progression free survival (PFS) after ASCT2
* Depth of best response (stable disease (SD), partial response (PR), very good partial response (VGPR), complete remission (CR), stringent complete remission (sCR)) after ASCT2
* Median Overall survival after ASCT2
* Treatment related mortality rate at ASCT2
* Mean duration of neutropenia (ANC < 0,5) at ASCT2
* Mean time until engraftment
* Mean duration of hospitalization after stem cell infusion at ASCT2
* The frequency of all serious adverse events according to version 5.0 of National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) during hospitalization and until day +100 after ASCT2.

Prespecified subgroups will include depth of best response prior to ASCT2, any specific maintenance therapies following ASCT2, patients receiving Granulocyte Colony Stimulating Factor (G-CSF) following ASCT, and patients receiving daratumumab as a part of induction or maintenance therapy at ASCT2.

In addition, an exploratory subgroup analysis is planned for patients with high-risk cytogenetics including p53-aberrations and patients with early relapse after ASCT1 (less than 3 years), although missing data is expected to be high.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of first relapse after previous ASCT for multiple myeloma according to the International Myeloma Working Group.
* Treated with a second ASCT (ASCT2) as part of second line treatment at UUH.
* Conditioning at ASCT2 with bortezomib-bendamustine-melphalan or high-dose melphalan only.

Exclusion Criteria:

* Double (tandem) ASCT in first or second line treatment
* Allogenic haematopoietic stem cell transplantation as part of first or second line therapy
* Failure to meet the minimal dataset, defined as: (date of ASCT1 and ASCT2, date of start of induction treatment for relapsed myeloma prior to ASCT2, medical records from hospitalization for ASCT2, at least one follow-up visit (unless early death before first follow-up visit), date of progression and first treatment of relapsed multiple myeloma after ASCT2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifty consecutive patients, who were referred to UUH for a second ASCT after relapse in multiple myeloma following HDM and ASCT between 1 Nov 2011 and 30 Jun 2018 and who received conditioning with bortezomib-bendamustine-melphalan will be included in this study. As a control group, 25 consecutive patients who were treated with HDM prior to 1 Nov 2011 and 25 consecutive patients following 30 Jun 2018. The patients will be identified through the local European Society for Blood and Marrow Transplantation (EBMT) registry at UUH.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-24 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Mean difference in time to next treatment (TNT) after ASCT1 and ASCT2 for each individual patient | 0.2-18 years
  Average time to next myeloma treatment within each individual patient making each patient as its' own control

SECONDARY OUTCOMES:
Median time to next treatment after ASCT2 | 0-18 years
  Time to start of next myeloma treatment after ASCT2
Median progression free survival (PFS) after ASCT2 | 0-18 years
  Time to progression or death after ASCT2
Median overall survival after ASCT2 | 0-18 years
  Survival until death from any cause
Depth of best response after ASCT2 | 0-24 months
  Best result after given treatment for myeloma
Treatment related mortality | 0-12 months
  Death due to any transplantation-related cause other than disease progression.
Mean duration of neutropenia at ASCT2 | 7-50 days
  Absolute neutrophil count (ANC) <0.5 x10^9
Mean time until engraftment at ASCT2 | 5-50 days
  Days from ASCT until ANC of 0.5 x 109/L or higher and total platelet count of 20 x 109/L and rising, without transfusion of thrombocytes.
Mean duration of hospitalization at ASCT2 | 7-50 days
  Days from ASCT until discharge
Frequency of severe adverse events at ASCT2 | 100 days
  All serious adverse events according to version 5.0 of National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) during hospitalization and until day +100 after ASCT2.

CONTACTS AND LOCATIONS:
Overall Officials: Honar Cherif, MD, PhD, Principal Investigator — Uppsala University
Locations (1):
- Akademiska sjukhuset, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, (text, tables, figures and appendices), will be available together with the study protocol after de-identification beginning 9 months and ending 5 years following article publication to researchers who provide a methodologically sound proposal. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: from 9 months after published article until 5 years.
Access Criteria: Researchers who provide a methodologically sound proposal. To gain access, data requestors will need to sign a data access agreement.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-26): https://cdn.clinicaltrials.gov/large-docs/29/NCT06245629/Prot_SAP_000.pdf